CLINICAL TRIAL: NCT01541722
Title: Oxidative Stress, Inflammation and Acute Decompensation in Urea Cycle Disorders
Status: Terminated | Type: Observational
Why Stopped: DSMB suggested closure due to low enrollment
Sponsor: Mark Batshaw (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor-Investigator, Mark Batshaw, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: RDCRN 5109; U54HD061221 (NIH)
Record Dates: First submitted 2012-02-08; First posted 2012-03-01 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Urea Cycle Disorders
Keywords: Urea cycle disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of the proposed study is to characterize the oxidative stress and inflammatory cytokine status in UCD during baseline and decompensated states.

DETAILED DESCRIPTION:
Protein turnover is a cyclic process with a net loss of protein in the fasting state and a net gain in the fed state contributing to nitrogen balance. These physiologic processes are impacted during infection; whole-body protein catabolism exceeds protein synthesis, resulting in net loss of whole-body protein. Patients with urea cycle disorders suffer episodes of periodic hyperammonemic crisis, often in association with intercurrent infections. The immediate cause of this decompensation is the increase in endogenous protein catabolism that is the endpoint of a cascade triggered by intercurrent illness. This increase in protein catabolism leads to elevations of serum amino acids and ammonia production, which cannot be eliminated by a dysfunctional urea cycle.

It is well known that infectious illnesses play a significant role in precipitating metabolic crises in urea cycle defects, presumably by triggering a cascade of events involving the release of inflammatory cytokines that lead to increased protein catabolism. Cytokines have also been implicated as distant mediators of oxidative stress. However, the correlation between oxidative stress, cytokine levels, and severity of a crisis is currently unclear.

The primary purpose of the proposed study is to characterize the oxidative stress and inflammatory cytokine status in UCD during baseline and decompensated states. The investigators will undertake measurements of selected markers of oxidative stress and cytokines in serum and urine during baseline and decompensated states in subjects with UCD in order to establish their prognostic value as biomarkers for disease severity and/or predictors of metabolic decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or highly-likely diagnosis of one of the eight UCDs as established for the Longitudinal Study (5101) (See section 4.2 Inclusion Criteria, Table 4 for diagnostic criteria for patients with UCD)
* Enrolled in Longitudinal Study of Urea Cycle Disorders (RDCRN UCDC #5101)

Exclusion Criteria:

* UCD patients who have undergone orthotopic liver transplantation
* Significant chronic medical co-morbidity that might confound the analysis as determined by the site investigators.
* Significant co-morbidities include but are not limited to:

  * diabetes, liver failure + cirrhosis
  * renal failure
  * cardiac disease
  * chronic inflammatory diseases
  * asthma requiring daily long-term control medications
  * significant respiratory disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Urea cycle disorders Inherited metabolic disorders N-acetylglutamate synthase (NAGS) deficiency Carbamyl phosphate synthetase I (CPSI) deficiency Ornithine transcarbamylase (OTC) deficiency Argininosuccinate synthetase (AS) deficiency (Citrullinemia) Argininosuccinate lyase (AL) deficiency (argininosuccinic aciduria Arginase (ARG) deficiency (hyperargininemia) Hyperornithinemia, hyperammonemia and homocitrullinuria (HHH) syndrome, or mitochondrial ornithine carrier (ORNT) deficiency Citrullinemia type II, mitochondrial aspartate/glutamate carrier (CITR) deficiency
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Laboratory values indicating oxidative stress | Change from baseline to period of decompensation up to one year
  Laboratory values that indicate oxidative stress include IL-1, IL-2, IL-6, and IL-8. These values will be analyzed as a panel (not individually) comparing baseline values to values during periods of decompensation.

CONTACTS AND LOCATIONS:
Overall Officials: George Diaz, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (11):
- United States (10):
  - University of California, Los Angeles, Los Angeles, California
  - The Children's Hospital, Aurora, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Case Western Medical College, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada